CLINICAL TRIAL: NCT03447795
Title: Alveolar Ridge Preservation Using Autogenous Tooth Graft Versus Autogenous Demineralized Dentin Graft. A Randomized Controlled Clinical Trial.
Brief Title: Alveolar Ridge Preservation Using Autogenous Tooth Graft Versus Autogenous Demineralized Dentin Graft.
Acronym: ARP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed AbdelRaouf Hussein, Dr. Ahmed Elfana, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19|01|02
Record Dates: First submitted 2018-02-15; First posted 2018-02-27 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Alveolar Ridge Preservation; Dentin Graft; Autogenous Tooth Bone Graft

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial (RCT) with parallel group, two arm, with 1:1 allocation ratio.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autogenous tooth grafted sites (Experimental)
  Interventions: Procedure: Alveolar ridge preservation
- autogenous demineralised dentin grafted sites (Active Comparator)
  Interventions: Procedure: Alveolar ridge preservation

INTERVENTIONS:
Procedure: Alveolar ridge preservation — grafting procedure using autogenous tooth.
  Other Names: ARP

SUMMARY:
Alveolar bone resorption following tooth extraction is unavoidable. Graft placement following extraction is recommended when considering restorative procedures afterwards. The extracted tooth was considered a clinical waste. However, it is now seen as a convenient and available source for graft material. Different protocols are applied to process the extracted tooth for obtaining the graft material and investigations are needed to assess the protocol with the best outcome.

DETAILED DESCRIPTION:
Autogenous graft is widely accepted as the gold standard for grafting procedures(Sakkas et al. 2017). And since the introduction of autogenous dentin graft for alveolar ridge preservation by Kim et al. clinically (Y.-K. Kim et al. 2010), it has increasingly attracted attention and teeth are no longer seen only as a waste. Tooth dentin has a chemical composition similar to that of alveolar bone; the inorganic content is 70%-75%, organic content 20%, and water content 10%, whereas alveolar bone has proportions of 65%, 25%, and 10% respectively(Y.-K. Kim et al. 2013). The similarity in chemical composition between dentin and alveolar bone, as well as its content of growth factors such as bone morphogenetic proteins (BMPs), made the dentin a successful graft for filing alveolar bone defects of same patient(Y.-K. Kim et al. 2010, Nampo et al. 2010, Y.-K. Kim et al. 2013) .

The technique proposed by Kim et al includes demineralization of the dentin as it reduces minerals content, exposes collagen fibrils and increases BMPs released thus promoting the process of osteogenesis(Y.-K. Kim et al. 2010). However, demineralisation step is time-consuming, taking several days, which challenges same visit application. As a result, two main approaches have been developed to overcome this obstacle. One approach is to maintain the demineralization step but with improving the technique to shorten the processing time(MURATA et al. 2010, E.-S. Kim 2015, Kabir et al. 2015). On the other hand, many investigators have used the whole tooth without demineralization and reported satisfactory clinical outcome(Gideon Hallel et al. 2014, Valdec et al. 2017). Hence, more investigations are needed to evaluate the technique with the best outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-restorable non-molar teeth
* Patients > 18 years old
* Motivated patients who are willing to continue the follow-up period

Exclusion Criteria:

* Compromised alveolar socket that is not contained to support graft material
* smokers and alcoholic patients.
* Patients with systemic conditions that may compromise hard tissue healing (i.e. poorly controlled diabetes, autoimmune diseases).
* Local infection at the site of extraction.
* Teeth with root canal filling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Cone beam computed tomography (CBCT) analysis | immediately and after 6 months of grafting
  CBCT scans will be taken at first day and at 6 months after the grafting procedures. The scans will be compared using predetermined reference points, buccolingual and vertical dimensions will be measured in cross-sectional images using the same reference points and lines. The difference in mm will be subtracted.

SECONDARY OUTCOMES:
Histological analysis | after 6 months of grafting
  Bone samples from at least one control and one intervention site will be taken during implant placement. Patients will be asked to sign and additional informed consent. A trephine bur will be used to obtain samples and then sent to the department of oral histology for assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided